CLINICAL TRIAL: NCT01397682
Title: Epidemiological Observatory on the Health Conditions of Inpatients Aged 65 or Older at the INRCA Research Hospitals
Acronym: report-AGE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA-01-2011
Record Dates: First submitted 2011-07-06; First posted 2011-07-19 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Aging; Inpatients
Keywords: Comprehensive Geriatric Assessment; Frail elderly; Italy/epidemiology; Geriatric Health Service; Polypharmacy; Biological Markers; Epidemiologic Research Design

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — plasma, serum, whole blood

INTERVENTIONS:
Other: blood sample collection — A blood sample will be drawn within 24 hours from admission for determination of biomarkers and genetic analyses

SUMMARY:
The goal of this research study is to collect clinical data, comprehensive geriatric assessment, risk factors, biological data and blood samples from inpatients aged 65 and older at the INRCA research hospitals (Italy). All data will be stored in a research bank and used to better clarify the mechanisms underlying the condition of "frailty" in aged patients. The database will be created on the INRCA server platform by establishing a safe HTTPS protocol.

DETAILED DESCRIPTION:
Life expectancy is continuously increasing in Italy. Aging is generally linked to adaptive modifications of organs and systems that reduce the functional reserve and increase the vulnerability to disease and addiction. This framework constitutes the condition of "frailty", which is associated to an increased risk of multiple adverse events as falls, fractures, disability, institutionalisation and death. To reduce the burden of disability and diseases affecting the quality of life of the elderly and, at the same time weighs heavily on health costs, a high level of managerial efficiency has to be achieved, planning the necessary health and care services and implementing measures to prevent disability in the fragile elderly. Indeed a strongly expanding area of gerontological and geriatric research is focusing on successful aging, that is characterised by a low probability of diseases and related disabilities, by a high level of physical and cognitive functionality and by an active social involvement in daily life. For this reason the project is based on the implementation of a validated system of comprehensive geriatric assessment able to provide detailed measures of the different possible interactions among risk factors. The study aimed at the descriptive-epidemiological collection of the health conditions of older in-patients at the different INRCA research hospitals (Italy). The data set will include personal data, information from the comprehensive geriatric assessment, clinical-care, biological and diagnostic data, collected routinely as well as ad hoc during hospitalisation. Moreover, a blood sample will be taken to performing biomarkers and genetic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* Inpatients at the different INRCA research hospital facilities (Italy)

Exclusion Criteria:

* Inpatients who have not/for those the informed consent was not given

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Inpatients aged 65 or older at the INRCA research hospital facilities of Ancona, Fermo, Casatenovo, Roma, Cosenza (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 2011-05-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Descriptive-epidemiological analysis of health conditions | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Collection of a set of data and indicators of the health conditions including personal data, clinical-care, biological and diagnostic data, treatments/procedures and drug therapy.

SECONDARY OUTCOMES:
Comprehensive geriatric assessment by INTERRAI-MDS-AC/VAOR-AC instrument | within 24 hours from admission and within 24 hours prior to discharge
  identification information, personal data at admission, assessment date, cognitive function, communication and vision, mood and behaviour, physical function, incontinence, diagnosis of the disease, health conditions, oral and nutrition status, skin conditions, medications, treatment and procedures, advanced directives, discharge potential, discharge, assessment information, anamnestic-clinical data, standardised clinical assessment, physical performance tests
Assessment of the functional capacities through specific performance tests | within 24 hours from admission and within 24 hours prior to discharge
  walking test, steps test, "chair standing", hand grip, articular extrusion
Evaluation of drugs consumption | within 24 hours from admission, during hospital stay and at discharge
  Drugs prior to admission, Drugs administered during hospital stay, Prescribed drugs at discharge
Identification of biomarkers: urinary markers of prostate disease | blood and urine samples drawn within 24 hours from admission
  score PCA3mRNA/PSAmRNA
Identification of biomarkers: immunological parameters | blood sample drawn within 24 hours from admission
  Leukocyte populations phenotype, Natural Killer activity in samples of leucocytes by means of citofluorimetric analysis
Identification of biomarkers: nutritional profile regarding trace elements | blood sample drawn within 24 hours from admission
  Identification of trace elements (Zn, Cu, Fe, Se) and alleles of genes that express proteins involved in their homeostasis (MT1A)
Identification of biomarkers: inflammation, oxidative stress and endothelial dysfunction | blood sample drawn within 24 hours from admission
  parameters of inflammation (pro- and anti-inflammatory cytokines: IL-6, IL-1, TNF-alpha, IL-10, IL-2, IL-17, IL-8; pro- and anti-inflammatory chemokines: MCP-1 and RANTES), parameters of oxidative stress (plasma total antioxidant capacity, determination of catalase, glutathione peroxidase, superoxide dismutase), and parameters of endothelial dysfunction (ADMA, SDMA, L-arginine, PAI-1)
Genetic analyses | blood sample drawn within 24 hours from admission
  assessment of: plasmatic and cellular (leukocytes) microRNA, mitochondrial DNA polymorphisms, length of telomeres of circulating leucocytes polymorphisms, epigenetic modifications of DNA in circulating leukocytes
Genomic wide testing | blood sample drawn within 24 hours from admission
  Genotyping by Affymetrix Genome-wide Human SNP array 6.0 will be performed by the Birdseed genotype calling algorithm, embedded in the Affymetrix Genotyping Console Software AGCS (Affymetrix), which is available at the Coordinating Center (INRCA).

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - INRCA Research Hospital, Ancona
  - INRCA Research Hospital, Casatenovo
  - INRCA Research Hospital, Cosenza
  - INRCA Research Hospital, Fermo

REFERENCES:
- [Background] Besdine RW, Wetle TF. Improving health for elderly people: an international health promotion and disease prevention agenda. Aging Clin Exp Res. 2010 Jun;22(3):219-30. doi: 10.1007/BF03324800. PMID 20634645
- [Derived] Di Rosa M, Sabbatinelli J, Soraci L, Corsonello A, Bonfigli AR, Cherubini A, Sarzani R, Antonicelli R, Pelliccioni G, Galeazzi R, Marchegiani F, Iuorio S, Colombo D, Burattini M, Lattanzio F, Olivieri F. Neutrophil-to-lymphocyte ratio (NLR) predicts mortality in hospitalized geriatric patients independent of the admission diagnosis: a multicenter prospective cohort study. J Transl Med. 2023 Nov 21;21(1):835. doi: 10.1186/s12967-023-04717-z. PMID 37990223
- [Derived] Corsonello A, Soraci L, Di Rosa M, Bustacchini S, Bonfigli AR, Lisa R, Liperoti R, Tettamanti M, Cherubini A, Antonicelli R, Pelliccioni G, Postacchini D, Lattanzio F. Prognostic Interplay of Functional Status and Multimorbidity Among Older Patients Discharged From Hospital. J Am Med Dir Assoc. 2022 Mar;23(3):499-506.e1. doi: 10.1016/j.jamda.2021.07.012. Epub 2021 Aug 9. PMID 34384766
- [Derived] Gagliardi C, Corsonello A, Di Rosa M, Fabbietti P, Cherubini A, Mercante O, Mazzei B, Postacchini D, Deales A, Bustacchini S, Lattanzio F. Preadmission Functional Decline Predicts Functional Improvement Among Older Patients Admitted to Acute Care Hospital. J Gerontol A Biol Sci Med Sci. 2018 Sep 11;73(10):1363-1369. doi: 10.1093/gerona/glx211. PMID 29087448
- [Derived] Bustacchini S, Abbatecola AM, Bonfigli AR, Chiatti C, Corsonello A, Di Stefano G, Galeazzi R, Fabbietti P, Lisa R, Guffanti EE, Provinciali M, Lattanzio F; Report-Age study group. The Report-AGE project: a permanent epidemiological observatory to identify clinical and biological markers of health outcomes in elderly hospitalized patients in Italy. Aging Clin Exp Res. 2015 Dec;27(6):893-901. doi: 10.1007/s40520-015-0350-3. Epub 2015 Mar 26. PMID 25809054